CLINICAL TRIAL: NCT05345041
Title: Keep it Movin': A Church-based Intervention to Improve Physical Function
Brief Title: Church-based Intervention to Improve Physical Function
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Elizabeth Lynch, Principal Investigator, Rush University Medical Center
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 21061405
Record Dates: First submitted 2022-04-15; First posted 2022-04-25 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Physical Function; Multiple Chronic Conditions
MeSH Terms: conditions — Multiple Chronic Conditions

STUDY DESIGN:
Intervention Model Description: The proposed study is a 12-month multi-level behavioral cluster randomized trial testing a church-based intervention to improve physical function (PF) in Americans with PF limitations (short physical performance battery [SPPB]<10). Churches in both arms (12 in each) will receive a virtual church-wide walking program which will be open to all church members, providing support for physical activity (PA) at interpersonal and community-levels. Churches will be randomized to either the church-wide walking program plus Keep it Movin' (KIM) intervention (intervention arm) or the church-wide walking program plus education (control arm). Using an active comparator will allow the assessment of whether the KIM intervention is more effective than a church-wide walking program along with improving PA individuals with PF limitations.
  Individuals who meet study inclusion criteria, including limited PF and at least two chronic conditions will be recruited from churches in both arms.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Keep it Movin' (Experimental)
  Interventions: Behavioral: Keep it Movin'
- Go 4 Life Self Guided Education (Active Comparator)
  Interventions: Behavioral: Go 4 Life Self Guided Education

INTERVENTIONS:
Behavioral: Keep it Movin' — Individual participants in churches randomized to the intervention arm will participate in the Keep it Movin' multi-component PA education program, as well as be encouraged by their church and study interventionist to participate in the church-wide walking program. Individuals enrolled in Keep It Movin' will attend weekly 90-minute sessions for 24 weeks. All sessions will include the structured physical activity component from the LIFE study intervention, with the following components, which were added to address needs of the target community: functional education, social support and problem-solving. To increase the functional gains seen in the LIFE pilot study and add content addressing self-management and PA with multiple chronic conditions (MCCs), the number of sessions in the proposed trial has been increased from 16 to 24 weeks.
  Arms: Keep it Movin'
Behavioral: Go 4 Life Self Guided Education — Individual participants in churches randomized to the comparator arm will receive the church-wide walking program and the Go4Life Your Everyday Guide to Exercise and Physical Activity which was developed by the National Institutes of Health National Institute on Aging to promote physical activity in older adults. This includes an evidence-based exercise guide and motivational tips to help older adults start and sustain an exercise program. The Go4Life guide will add individual level education and encouragement to the interpersonal and community levels of intervention provided by the church-wide walking program.
  Arms: Go 4 Life Self Guided Education

SUMMARY:
This is a 12-month multi-level behavioral cluster randomized trial testing a church-based intervention to improve physical function (PF) in Americans with PF limitations.

ELIGIBILITY:
Inclusion Criteria:

Churches (Community-level):

* Membership of 300 or more adults
* Located in Cook, Lake, Dupage, Will, McHenry, Kane, or Kendall counties

Participants (Individual-level):

* Age 40 or older
* Have mobility limitations (defined as SPPB score of ≤9)
* Ambulatory, defined as able to get out of a chair and walk without assistance without using a straight cane
* Able to speak and read English
* Attend recruitment church; and
* Safe to begin an exercise program, which will be determined using the Exercise Assessment and Screening for You (EASY) Tool.

Exclusion Criteria:

Participants (Individual-level):

* Severe cognitive impairment, defined as five or more errors on the Short-Portable Mental Status Questionnaire
* Unable to consistently attend group classes at a scheduled time due to lack of reliable transportation, schedule conflicts, travel, plans to relocate, upcoming surgery, etc.
* Participating in a medically supervised rehabilitation program such as cardiac rehab
* Inpatient treatment for a psychiatric condition within the past 6 months, or currently receiving treatment for schizophrenia or other serious psychiatric illness
* Contraindications to exercise determined using the EASY/healthcare follow-up
* Congestive heart failure New York Health Association (NYHA) Class I or higher; unstable angina; heart attack or stroke within past 6 months
* Visual or hearing impairment.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Physical Function | Measured at baseline and 6 months and 12 months after start of the intervention
  Objective physical function will be measured using the Short Physical Performance Battery (SPPB) an instrument commonly used to measure physical performance within the aging population.

SECONDARY OUTCOMES:
Change in Physical Activity | Measured at baseline and 6 months and 12 months after start of the intervention
  Objective physical activity (i.e., time spent in moderate and vigorous physical activity) will be collected via a wrist worn accelerometer (ActiGraph GT9X Link activity monitor) collected over 4-7 days. The ActiGraph GT9X Link provides physical activity data including raw acceleration, energy expenditure, steps taken, physical activity intensity, activity and sedentary bouts, and heart rate intervals.
Change in Self-Reported Physical Activity | Measured at baseline and 6 months and 12 months after start of the intervention
  Self reported physical activity will be evaluated using the Community Healthy Activities Model Program For Seniors (CHAMPS) questionnaire. The CHAMPS physical activity questionnaire is designed to promote physical activity in seniors. The CHAMPS tool is a 41-item questionnaire that asks about the length of time spent doing certain activities (less than an hour to 9 or more hours) in the past 4 weeks.
Change in Self-Reported Physical Function | Measured at baseline and 6 months and 12 months after start of the intervention
  Self-report of physical function will be evaluated by the Functional Status Questionnaire. The survey is a geriatric tool designed for participants to self-report capturing the participants' physical, psychological, social and role functions.
Change in Social Support | Measured at baseline and 6 months and 12 months after start of the intervention
  Social support for exercise will be measured using the Social Support & Exercise Survey Self-efficacy questionnaire.
Change in Quality of Life | Measured at baseline and 6 months and 12 months after start of the intervention
  Quality of life will be measured using EuroQual (EQ-5D-5L) questionnaire. The measure evaluates the participant's perception of their "health today" with respect to mobility, self-care, usual activities, pain/discomfort, and anxiety depression. the items are evaluated on a 5-point scale ranging from "no problem" in the area to "extreme problem" in the area.
Change in Self-efficacy | Measured at baseline and 6 months and 12 months after start of the intervention
  Self efficacy will be measured using The Self-Efficacy for Exercise Scale consisting of 9 hypothetical situations like weather, boredom that could impact a person's ability to exercise.

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

DOCUMENTS (1):
  • Informed Consent Form (2023-04-13): https://cdn.clinicaltrials.gov/large-docs/41/NCT05345041/ICF_000.pdf